CLINICAL TRIAL: NCT07331363
Title: Evaluation of the Effect of Using Ultrasound Robots for Breast Cancer Screening: A Multicenter, Parallel-group, Cluster Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaoxv Yin, PhD, Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HuazhongU20251203
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Ultrasound
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: Using an ultrasound robot to screen the subjects (Experimental)
  Interventions: Device: Screening of the subjects was conducted using an ultrasonic robot.
- The subjects are scanned with traditional hand-held ultrasound. (No Intervention): The subjects are scanned with traditional hand-held ultrasound.The images are diagnosed by radiologists.

INTERVENTIONS:
Device: Screening of the subjects was conducted using an ultrasonic robot. — The ultrasound robot automatically scans the breasts of subjects via its mechanical arm and generates images.The diagnosis is made based on the radiologist's interpretation of the images.
  Arms: Intervention group: Using an ultrasound robot to screen the subjects

SUMMARY:
The goal of this clinical trial is to learn if robotic ultrasound screening works as well as or better than traditional sonographer-led screening for detecting breast cancer. It will also explore how well participants follow recommended post-screening care. The main questions it aims to answer are:

Does robotic ultrasound screening detect more cases of breast cancer compared to traditional sonographer-led screening? How well do participants follow up on recommended care after robotic ultrasound screening? Researchers will compare robotic ultrasound screening to traditional sonographer-led screening to see if robotic ultrasound works effectively for breast cancer screening.

Participants will:

Receive a breast ultrasound performed either by a robotic system or a human sonographer.

Undergo follow-up management based on their BI-RADS classification.

ELIGIBILITY:
Inclusion Criteria:

1. women aged 35-64 years
2. no history of breast cancer
3. ownership and ability to use a smartphone
4. willingness to participate in the screening program.

Exclusion Criteria:

1. Women who have undergone breast removal surgery;
2. Pregnant and lactating women;
3. Women who have undergone breast cancer screening within the past year;

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70000 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-12-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
The detection rate of breast cancer | After participating in the screening, the subjects will be followed up for 24 months.
  Number of detected ductal carcinoma in situ (DCIS) and invasive breast cancers divided by the total number of screened participants.

SECONDARY OUTCOMES:
Cancer type | After participating in the screening, the subjects will be followed up for 24 months.
  Non-invasive cancer (DCIS), early invasive cancer, and invasive cancer.
The early diagnosis rate | After participating in the screening, the subjects will be followed up for 24 months.
  The early diagnosis rate is defined as the number of breast cancer cases with TNM stage 0, I, or IIa divided by the number of women diagnosed with breast cancer or other malignant breast tumors during screening*100.
Lymph node status | After participating in the screening, the subjects will be followed up for 24 months.
  Presence of lymph node metastasis; size, morphology, internal structure, margin characteristics, and vascularity of metastatic lymph nodes.
Breast cancer clinical stage | After participating in the screening, the subjects will be followed up for 24 months.
  TNM staging, representing tumor size (T), lymph node involvement (N), and distant metastasis (M).
Histological Grading of Breast Cancer | After participating in the screening, the subjects will be followed up for 24 months.
  The internationally accepted Nottingham Histological Grading System is used. This system provides a semi-quantitative and objective assessment of invasive breast cancer. It evaluates three parameters: the proportion of tubule formation, nuclear pleomorphism, and mitotic count. The scores of the three parameters are added together. A total score of 3-5 indicates Grade 1 (G1, well-differentiated/low grade). A total score of 6-7 indicates Grade 2 (G2, moderately differentiated/intermediate grade). A total score of 8-9 indicates Grade 3 (G3, poorly differentiated/high grade).
Breast cancer screen recall rate | After participating in the screening, the subjects will be followed up for 24 months.
  Breast cancer screen recall is defined as further assessment triggered by abnormal ultrasound findings (BI-RADS 0 or 3 and above). The recall rate is the number of women actually recalled divided by the number of women screened.
The positive predictive value | After participating in the screening, the subjects will be followed up for 24 months.
  The positive predictive value of recall is the percentage of recalled women who are diagnosed with breast cancer.
The breast cancer biopsy rate | After participating in the screening, the subjects will be followed up for 24 months.
  The breast cancer biopsy rate is defined as the number of women who actually underwent biopsy divided by the number of women screened. The positive predictive value of biopsy is defined as the percentage of women diagnosed with breast cancer among those who received a biopsy.
Referral adherence rate | After participating in the screening, the subjects will be followed up for 24 months.
  Defined as the average adherence to recommended referral for confirmed diagnosis (biopsy and histopathology). It is calculated as the number of women actually referred divided by the number of women recommended for referral.
Interval cancer incidence | After participating in the screening, the subjects will be followed up for 24 months.
  Defined as the proportion of women who had a negative or false-positive screening (i.e., no ductal carcinoma in situ or invasive breast cancer) and were subsequently diagnosed with invasive breast cancer within a certain period after screening. Following the national breast cancer screening guideline recommending screening every 2-3 years, this study will evaluate the interval cancer incidence at 24 months, i.e., the proportion of women diagnosed with breast cancer 24 months after a negative screen or 6-24 months after a false-positive screen.
Breast cancer mortality | After participating in the screening, the subjects will be followed up for 24 months.
  Defined as the number of deaths due to breast cancer within 24 months after screening divided by the total number of women screened.
All-cause mortality | After participating in the screening, the subjects will be followed up for 24 months.
  Defined as the total number of deaths from any cause within 24 months after screening divided by the total number of women screened.
Post-screening management adherence | After participating in the screening, the subjects will be followed up for 24 months.
  Defined as the proportion of women who completed the recommended follow-up medical actions after screening (referral, re-examination, additional tests, etc.). The adherence rate is calculated as the number of participants who completed the recommended management within the specified time / the number of participants requiring further management * 100%.

CONTACTS AND LOCATIONS:
Locations (1):
- Rural health centers and community health centers, Xiantao, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided